CLINICAL TRIAL: NCT02461966
Title: Evaluation of the Role of Aflatoxin as an Environmental Risk Factor Attributable to Liver Cancer in Nile Delta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, sponsor investigator, Tanta University
Organization: Tanta University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Aflatoxin
Record Dates: First submitted 2015-05-31; First posted 2015-06-03 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — Aflatoxins

STUDY DESIGN:
Masking Description: No Masking
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hepatocellular carcinoma (HCC) (Other): Estimation of serum aflatoxin level in 40 patients with hepatocellular carcinoma (HCC)
  Interventions: Other: Aflatoxin
- 20 cirrhotic patients (Other): Estimation of serum aflatoxin level in 20 patients with liver cirrhosis
  Interventions: Other: Aflatoxin
- Control group (Other): Estimation of serum aflatoxin level in 15 individuals, as a control group in patient house whom share the same quality of life and whom were neither HCC patients nor cirrhotic patients, were invited to share in the study
  Interventions: Other: Aflatoxin

INTERVENTIONS:
Other: Aflatoxin — Evaluation of Aflatoxin level

SUMMARY:
Hepatocellular carcinoma is multifactorial in etiology and complex in pathogenesis, the blend of risk factors differs in different parts of the world, and this may explain in part the diverse biologic characteristics of HCC in different populations .

Exposure to aflatoxin is an additional risk factor for the development of HCC, through damage of DNA in liver cells and mutation in p53 tumor suppressor gene . A previous study showed that aflatoxin B1 has a considerable role in the development of HCC among Egyptians .

Clinical studies have shown that AFB1 selectively targets at the third base position of codon 249 of the human p53 gene, a known mutational hotspot in human hepatocellular carcinoma (HCC) . A significant association between aflatoxin exposure and HCC has been reported in hyperendemic areas . A synergistic interaction between AFB1 exposure and viral hepatitis B (HBV) infection on HCC risk has been reported in several epidemiologic studies.

Aflatoxin exposure may be associated with advanced liver disease in chronic hepatitis C (HCV) patients. Levels of AFB1-albumin/albumin were significantly related to ultrasono-graphic hepatic parenchyma scores in anti-HCV-positive subjects .

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common malignancy in the world and the third most common cause of cancer-related deaths complicating liver cirrhosis in most cases.

In Egypt, there has been a remarkable increase of the proportion of HCC among chronic liver diseases (CLD) patients from 4.0% to 7.2% over a decade. This rising proportion may be explained by the increasing risk factors such as the emergence of hepatitis C virus (HCV) over the same period of time, the contribution of hepatitis B virus (HBV) infection, improvement of the screening programs and diagnostic tools of HCC as well as the increased survival rate among patients with cirrhosis to allow time for some of them to develop HCC .

Hepatocellular carcinoma is multifactorial in etiology and complex in pathogenesis, the blend of risk factors differs in different parts of the world, and this may explain in part the diverse biologic characteristics of HCC in different populations .

Exposure to aflatoxin is an additional risk factor for the development of HCC, through damage of DNA in liver cells and mutation in p53 tumor suppressor gene . A previous study showed that aflatoxin B1 has a considerable role in the development of HCC among Egyptians .

Clinical studies have shown that AFB1 selectively targets at the third base position of codon 249 of the human p53 gene, a known mutational hotspot in human hepatocellular carcinoma (HCC) . A significant association between aflatoxin exposure and HCC has been reported in hyperendemic areas . A synergistic interaction between AFB1 exposure and viral hepatitis B (HBV) infection on HCC risk has been reported in several epidemiologic studies.

Aflatoxin exposure may be associated with advanced liver disease in chronic hepatitis C (HCV) patients. Levels of AFB1-albumin/albumin were significantly related to ultrasono-graphic hepatic parenchyma scores in anti-HCV-positive subjects .

ELIGIBILITY:
Inclusion Criteria:

* cirrhotic patient with and without HCC

Exclusion Criteria:

* Malignancy other than HCC

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sharaf-eldin, Prof, Principal Investigator — hepatology dept-Tanta; Raafat Salah, Professor, Study Director — hepatology dept-Tanta; hanan Soliman, Prof, Study Chair — hepatology dept-Tanta; Sherief abd-elsalm, lecturer, Study Chair — hepatology dept-Tanta; Walaa Elkhalawany, lecturer, Study Chair — hepatology dept-Tanta
Locations (1):
- Tanta university - faculty of medicine, Cairo, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Hepatocellular Carcinoma (HCC): Estimation of serum aflatoxin level in 160 patients with hepatocellular carcinoma (HCC)
  Aflatoxin: Evaluation of Aflatoxin level
- Cirrhotic Patients: Estimation of serum aflatoxin level in 80 patients with liver cirrhosis
  Aflatoxin: Evaluation of Aflatoxin level
- Control Group: Estimation of serum aflatoxin level in 60 individuals, as a control group in patient house whom share the same quality of life and whom were neither HCC patients nor cirrhotic patients, were invited to share in the study
  Aflatoxin: Evaluation of Aflatoxin level
Period: Overall Study
Arm/Group | Hepatocellular Carcinoma (HCC) | Cirrhotic Patients | Control Group
Started | 160 | 80 | 60
Completed | 160 | 80 | 60
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hepatocellular Carcinoma (HCC) | Cirrhotic Patients | Control Group | Total
Number analyzed (Participants) | 160 | 80 | 60 | 300
Age, Categorical [Count of Participants; unit: Participants] — Age, categorical numerical
  Participants
    <=18 years | 0 | 0 | 0 | 0
    Between 18 and 65 years | 132 | 63 | 39 | 234
    >=65 years | 28 | 17 | 21 | 66
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 58.58 (9.58) | 50.00 (8.72) | 27.80 (5.06) | 45 (23.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 24 | 24 | 76
  Male | 132 | 56 | 36 | 224
Region of Enrollment [Number; unit: participants]
  Egypt | 160 | 80 | 60 | 300

OUTCOME MEASURES:

1. Primary Outcome: Serum Aflatoxin Level in Liver Cancer Patients
Description: Serum aflatoxin level in liver cancer patients in comparison to liver cirrhosis and controls.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng\ml
Groups:
- 80 Cirrhotic Patients: Estimation of serum aflatoxin level in 80 patients with liver cirrhosis
  Aflatoxin: Evaluation of Aflatoxin level
Arm/Group | Hepatocellular Carcinoma (HCC) | 80 Cirrhotic Patients | Control Group
Number analyzed (Participants) | 160 | 80 | 60
ng\ml | 7.96 (2.06) | 6.10 (1.71) | 4.13 (1.67)

ADVERSE EVENTS:
Time Frame: 2 years
Description: 0 means no side effects
Arm/Group | Hepatocellular Carcinoma (HCC) | Cirrhotic Patients | Control Group
Serious Adverse Events (participants affected / at risk) | 0/160 | 0/80 | 0/60
Other Adverse Events (participants affected / at risk) | 0/160 | 0/80 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No